CLINICAL TRIAL: NCT01792557
Title: Crystallized Phenol Application Versus Transposition Flaps for Treatment of Sacrococcygeal Pilonidal Disease: A Prospective Randomized Study
Brief Title: Crystallized Phenol Versus Transposition Flaps for Treatment of Pilonidal Disease: A Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: S.B. Konya Education and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEAH06021301; U1111-1139-3538 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Pilonidal Sinus
Keywords: Pilonidal sinus; Crystallized phenol; Limberg Flap; Modified Limberg Flap; Karydakis; Recurrence; Complications; Recovery duration; Time to return to work
MeSH Terms: conditions — Pilonidal Sinus; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phenol (Active Comparator): Crystallized Phenol Group
  Interventions: Drug: Crystallized phenol
- Limberg (Active Comparator): Limberg Flap Group
  Interventions: Procedure: Limberg Flap
- Modified Limberg (Active Comparator): Modified Limberg Flap Group
  Interventions: Procedure: Modified Limberg Flap
- Karydakis (Active Comparator): Karydakis Flap Group
  Interventions: Procedure: Karydakis Flap

INTERVENTIONS:
Drug: Crystallized phenol — Crystallized phenol application for pilonidal disease treatment. After sacrococcygeal region of the patient is cleaned from hairs, hairs inside the sinus are removed than crystallized phenol is applied in to the cleaned sinus. Following 2 minutes of phenol exposure, crystallized phenol is removed from the sinus. Crystallized phenol application will be repeated weekly for 4 weeks.
  Arms: Phenol
Procedure: Limberg Flap — Limberg Flap surgery for pilonidal disease treatment
  Arms: Limberg
Procedure: Modified Limberg Flap — Limberg flap surgery rhomboid incision is made asymmetrically 2-3 cm lateral to the midline on the side opposite to the donor area.
  Arms: Modified Limberg
Procedure: Karydakis Flap — Karydakis Flap surgery for pilonidal disease treatment
  Arms: Karydakis

SUMMARY:
Although surgical techniques such as limberg flap. modified limberg flap and karydakis are currently most popular treatment methods for pilonidal disease, crystallized phenol application is also successfully used for pilonidal sinus treatment by different centers. We believe crystallized phenol application could become a good alternative to popular surgical interventions using transposition flaps.

DETAILED DESCRIPTION:
Pilonidal sinus disease (PSD) is usually located at sacrococcygeal region of the body and mostly effect young males causing loss of labor and school time. Its incidence is reported 26 per 100000 in a Norwegian study. Although there are many treatment modalities either surgical or conservative, ideal treatment is still a matter of debate. Surgical techniques such as limberg flap, modified limberg flap and karydakis are most popular treatment methods for pilonidal disease crystallized phenol application is also successfully used for pilonidal sinus treatment by different centers. We would like to compare flap techniques and crystallized phenol application for complications, recurrence, patient comfort, duration of recovery and return to work. We believe crystallized phenol application could become a good alternative to popular surgical interventions using transposition flaps.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pilonidal disease

Exclusion Criteria:

* Previous history of pilonidal disease treatment
* Pregnant or breast-feeding women
* Systemic diseases that would affect wound healing
* Diabetes
* Chronic renal failure
* Autoimmune diseases
* Malignant diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of recurrence | 3rd year
  Patients will be followed up for recurrence for three years. Total recurrence will be evaluated at the end of 3rd year.

SECONDARY OUTCOMES:
Assessment of patient comfort | 1st year
  Patients will be queried for patient comfort at the end of first year
Assessment of recovery duration | 3rd month
  Post procedure wound recovery duration will be recorded
Assessment of complications | 3rd month
  Patients will be followed up for procedure related complications.

OTHER OUTCOMES:
Assessment of time before patient returns to work/routine physical activity | 3rd month
  Patients will be queried for when they felt comfortable to return to work and/or their routine physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Doğru, M.D., Study Director — Konya Education and Research Hospital
Locations (1):
- Konya Education and Research Hospital, Meram, Konya, Turkey (Türkiye)

REFERENCES:
- [Background] Dogru O, Camci C, Aygen E, Girgin M, Topuz O. Pilonidal sinus treated with crystallized phenol: an eight-year experience. Dis Colon Rectum. 2004 Nov;47(11):1934-8. doi: 10.1007/s10350-004-0720-y. PMID 15622588
- [Background] Akin M, Leventoglu S, Mentes BB, Bostanci H, Gokbayir H, Kilic K, Ozdemir E, Ferahkose Z. Comparison of the classic Limberg flap and modified Limberg flap in the treatment of pilonidal sinus disease: a retrospective analysis of 416 patients. Surg Today. 2010 Aug;40(8):757-62. doi: 10.1007/s00595-008-4098-7. Epub 2010 Jul 30. PMID 20676861
- [Background] Keshava A, Young CJ, Rickard MJ, Sinclair G. Karydakis flap repair for sacrococcygeal pilonidal sinus disease: how important is technique? ANZ J Surg. 2007 Mar;77(3):181-3. doi: 10.1111/j.1445-2197.2006.04003.x. PMID 17305997
- [Background] Cihan A, Mentes BB, Tatlicioglu E, Ozmen S, Leventoglu S, Ucan BH. Modified Limberg flap reconstruction compares favourably with primary repair for pilonidal sinus surgery. ANZ J Surg. 2004 Apr;74(4):238-42. doi: 10.1111/j.1445-2197.2004.02951.x. PMID 15043735